CLINICAL TRIAL: NCT01523041
Title: A Randomised, Double Blind, Single Centre, Three Period Crossover Trial Testing the Bioequivalence of Two Formulations of Biphasic Insulin Aspart 70 and Characterising the Pharmacokinetics of Biphasic Insulin Aspart 50 in Healthy Male Subjects
Brief Title: Comparison of Two Formulations of Biphasic Insulin Aspart 70
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1144
Record Dates: First submitted 2012-01-25; First posted 2012-02-01 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- BIAsp 70 clinical trial formulation (Experimental)
  Interventions: Drug: biphasic insulin aspart 70
- BIAsp 70 final formulation (Experimental)
  Interventions: Drug: biphasic insulin aspart 70
- BIAsp 50 final formulation (Experimental)
  Interventions: Drug: biphasic insulin aspart 50

INTERVENTIONS:
Drug: biphasic insulin aspart 70 — A single dose administrated subcutaneously (s.c., under the skin)
  Arms: BIAsp 70 clinical trial formulation
Drug: biphasic insulin aspart 70 — A single dose administrated subcutaneously (s.c., under the skin)
  Arms: BIAsp 70 final formulation
Drug: biphasic insulin aspart 50 — A single dose administrated subcutaneously (s.c., under the skin)
  Arms: BIAsp 50 final formulation

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare two formulations of biphasic insulin aspart 70 and characterise the pharmacokinetics of biphasic insulin aspart 50 and biphasic insulin aspart 70 in healthy male subjects.

DETAILED DESCRIPTION:
Each subject participated in three treatment periods, and were randomly assigned to each of the six treatment sequences in varying order

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Considered generally healthy upon completion of medical history and physical examination as judged by the Investigator
* Body mass index (BMI) between 19-27 kg/m^2
* Fasting plasma glucose between 3.8-6.0 mmol/L

Exclusion Criteria:

* Participation in any other clinical trial involving other investigational products within the last three months
* Clinically significant abnormal haematology or biochemistry screening tests, as judged by the Investigator
* Any serious systemic infectious disease that occurred in the 4 weeks prior to the first dose of test drug

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1999-11-03 (Actual); Primary Completion 1999-11-30 (Actual); Study Completion 1999-11-30 (Actual)

PRIMARY OUTCOMES:
Area under the insulin aspart curve in the interval from 0-24 hours

SECONDARY OUTCOMES:
Cmax, maximum insulin aspart concentration
tmax, the time to maximum insulin aspart concentration
t½, terminal half-life
Cmin, minimum glucose concentration
tmin, time to minimum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Leeds, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com